CLINICAL TRIAL: NCT02935777
Title: Investigation of the Acute Effect of Pomegranate Extract on Cognitive Function in Human Volunteers: A Double-blind, Placebo-controlled, Crossover Trial
Brief Title: Acute Effect of Pomegranate Extract on Cognitive Function
Acronym: POM-03
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Angela Stockton (Other)
Collaborators: Northumbria University (Other)
Responsible Party: Sponsor-Investigator, Angela Stockton, PhD Researcher, Queen Margaret University
Organization: Queen Margaret University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: POM-03
Record Dates: First submitted 2016-10-06; First posted 2016-10-18 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Mental Processes
Keywords: Pomegranate extract; cognitive function; cognition; polyphenols; memory
MeSH Terms: interventions — pomegranate fruit rind

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pomegranate Extract (Experimental): POMANOX® pomegranate extract capsules with water by mouth, once. Dosage: 2 capsules
  Capsules weigh1.083g and contain: 210mg punicalagin, 328mg other pomegranate polyphenols (e.g. flavonoids and ellagic acid), 0.37mg anthocyanins and maltodextrin.
  Interventions: Dietary Supplement: Pomegranate Extract
- Placebo (Placebo Comparator): Identical placebo capsules by mouth, administered once. Dosage 2 capsules. Each capsule contains maltodextrin to provide PE capsule energy equivalent i.e.6.52 kcal or 27.28kJ.
  Interventions: Dietary Supplement: Placebo capsule

INTERVENTIONS:
Dietary Supplement: Pomegranate Extract — The first computer cognitive testing session lasting approximately 45 minutes is undertaken by participants. After completion, intervention capsules are administered. After a 60 minute absorption period, the cognitive testing session is re-administered.
  Other Names: POMANOX
  Arms: Pomegranate Extract
Dietary Supplement: Placebo capsule — One computer cognitive testing session lasting approximately 45 minutes is undertaken by participants. After completion, placebo capsules are administered. After a 60 minute absorption period, the cognitive testing session is re-administered.
  Arms: Placebo

SUMMARY:
The double-blinded, randomised, placebo-controlled crossover pilot study is conducted as a two week intervention after a pre-intervention registration and preparation period.

This study explores whether acute supplementation with pomegranate extract can modulate indicators of cognitive function and mood in healthy adults. Changes in physiological and biochemical markers are also investigated.

DETAILED DESCRIPTION:
Participants are asked to visit the QMU clinical lab three times. The first visit is for general information, form completion, measurements and consent plus a practise session on COMPASS, the study computer software. Information and consent forms and a screening questionnaire are completed. Basic information such as age, sex, weight, height and blood pressure data are recorded. Lab visits 2 and 3, which are a week apart, constitute the intervention phase.

Participants are randomly assigned to either the pomegranate extract (PE) or placebo group.The researcher and participants are blinded to which capsules they are taking until data collection is complete. The randomisation process is carried out by independent technical staff who use an internet random number generator site to allocate treatment. The PE and placebo capsules look identical and are placed in sealed, labeled, pre-prepared opaque containers numbered by technicians.

At the next lab session (visit 2) participants begin their randomised study arm, taking either two pomegranate extract or two placebo capsules with water by mouth. Participants repeat the procedure at visit 3, where they crossover to the remaining intervention. Thus if participant A consumed placebo capsules at visit 2, the participant would take pomegranate extract capsules at visit 3, following a washout period of a week. If participant B consumed pomegranate extract on visit 2, the participant would then take the placebo capsules at visit 3.

At each visit, participants complete two computer testing sessions lasting approximately 45 minutes - one pre and one post capsule ingestion. After the capsule is taken there is a one hour absorption period before the next computer test session begins.

Participants are fasted from tea and coffee overnight and abstain for the period of the intervention in the morning. On the day before the tests, they are requested to refrain from alcohol, recreational drugs, and vigorous exercise.

Participants are also required to restrict herbal extracts, food supplements and polyphenols such as dark chocolate, fruit rich in polyphenols and antioxidants to less than three portions for 24 hrs beforehand. A 24 hour pre test food diary is completed to assist in compliance. Participants are also advised to have a good night's sleep - at least 6-8 h during the night before the study day - and should not be more stressed than usual. These aspects are confirmed before participants are allowed to commence their sessions.

Pre-study saliva collection is completed at home by participants early in the morning. This provides a biochemical marker which aims to support both cognitive findings and the results from the Bond Lader mood questionnaire completed during the computer testing. Instructions are given to participants for saliva collection and the samples analysed for cortisol and cortisone. Participants are instructed to have their usual breakfast except for coffee or tea. Blood pressure is taken pre and post study on visits 2 and 3.

The baseline computerised cognitive test battery is administered in the clinic at 9am lasting around 45 mins. The investigator then observes the participants consuming their scheduled capsules. After a one hour quiet absorption period around 11am, blood pressure is taken again. The post cognitive testing battery is completed once more and then a second post study saliva collection is taken. Participants complete the intervention around 12 noon. All assessments are carried out on a QMU computer, with the same laptop used by each participant at baseline and post intervention assessments.

The cognitive testing is conducted under controlled laboratory conditions with the assessments at baseline and post study always performed at the same time of day (between 0830 and 1200) for each participant.

Participant responses to the cognitive tests are recorded automatically by the computer software during the testing battery at visits 2 and 3.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Aged 18-65
* Enjoy computer tasks

Exclusion Criteria:

* Diagnosis with any neurological, psychiatric or significant medical condition which could affect cognitive function
* Known cognitive impairment
* Use of any prescription, herbal or recreational drugs
* Gastrointestinal disease
* Pregnancy or breastfeeding
* Pomegranate allergy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04; Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Simple reaction time (attention and vigilance, speed of attention) | 1-2 hours
  Reaction time in msec.
Choice reaction time (attention and vigilance, speed and accuracy of attention) | 1-2 hours
  Arrows pointing left and right will appear on the screen at irregular intervals. The participant is required to indicate the direction of the arrow as quickly as possible, whenever an arrow is displayed. Measured by % accuracy, overall correct responses and reaction time (ms).
Bond Lader mood scales | 1-2 hours
  Mood is measured via the Bond Lader series of mood scales, each scored out of 100. From these scales three composite scores are calculated describing feelings of 'Alert', 'Calm' and 'Content', also presented as a score out of 100.
Digit vigilance (attention and vigilance, speed and accuracy of attention) | 1-2 hours
  A fixed number will appear on the right of the screen and a series of changing numbers will appear on the left side of the screen. Participants are required to make a response when the number on the left matches the number on the right. Measured by reaction time (ms) and %accuracy of responses.
Word presentation (secondary memory) then delayed Word recall (quality of memory) | 1-2 hours
  A list of words is displayed on the screen, one word at a time. Participants are given 60 seconds to write down as many of the words they were shown earlier as they can. This task was performed following following a delay between the presentation and recall (delayed recall). no of correct responses and % accuracy.
Word recognition (secondary memory, quality and speed of memory) | 1-2 hours
  All target words that were shown during Word Presentation plus an equal number of decoys will be displayed on the screen one at a time. Participants indicate if they remember seeing the word earlier or not. measured by correct no of responses, errors and reaction time (ms).
Rapid Visual Information Processing (RVIP) (cognitive demand) | 1-2 hours
  A series of numbers are displayed individually on the screen in quick succession (at a rate of 100 numbers per minute) and participants are required to respond when they see 3 odd numbers in a row or three even numbers in a row. Measured by % accuracy, no of false alarms and reaction time (ms).
Picture presentation (secondary memory) and delayed recognition(secondary memory, speed and quality of memory) | 1-2 hours
  A series of pictures are displayed on the screen, one at a time. After a delay, all target pictures shown during Picture Presentation plus an equal number of decoys will be displayed on the screen one at a time. For each stimulus participants select 'Yes' or 'No' to indicate if they have seen the picture before or not. The task is measured by reaction time (ms), % accuracy and no of correct responses.
Corsi blocks lite (working memory, spatial memory) | 1-2 hours
  Blue squares on a black background are displayed on the screen. Some of them change to red and back to blue again in a sequence. Participants are required to remember this sequence. The task is repeated five times at each level of difficulty with the sequence span increasing from 4 upwards, until the participant can no longer correctly recall the sequences. The task continues up to 6 squares in each sequence, while participants make enough correct responses. As soon as they make less than 3 correct responses (out of the five in one level) the task will end. All participants complete levels 4-6 regardless of incorrect responses. Results are measured by a span score: This score is calculated as the average of the last 3 correctly completed trials. For example, if the participant correctly responds to all five Level 4 trials and only one Level 5 trial, their span score would be 4.3 [(4 + 4 + 5)/3].

SECONDARY OUTCOMES:
Pre and post blood pressure changes | 1-2 hours
  Measurement of systolic and diastolic blood pressure in mmHg.
Pre-post cortisol and cortisone changes | 3-4 hours
  Collection of saliva which is processed via ELISA to measure cortisol and cortisone in ng/mL

CONTACTS AND LOCATIONS:
Overall Officials: Emad Aldujaili, Study Director — Dean of Pharmacy, Jordan University
Locations (1):
- Queen Margaret University, Edinburgh, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No